CLINICAL TRIAL: NCT07282561
Title: Role of Nutritional Status in Functional Recovery of Older Adults Undergoing Virtual Reality-augmented Shoulder Rehabilitation (VIR)
Acronym: VIR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Claudio Pedone (Other)
Responsible Party: Sponsor-Investigator, Claudio Pedone, Professor, Fondazione Policlinico Universitario Campus Bio-Medico
Organization: Fondazione Policlinico Universitario Campus Bio-Medico (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 37.25_CET2_CBM_VIR; PNC0000007 - "Fit4MedRob" (Other Grant/Funding Number: Ministero dell'Università e della Ricerca)
Record Dates: First submitted 2025-11-17; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-11

CONDITIONS: Shoulder Arthroplasty; Rehabilitation; Virtual Reality; Malnutrition Elderly

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality-augmented shoulder rehabilitation (Active Comparator)
  Interventions: Device: Oculus Quest
- Usual care (No Intervention)

INTERVENTIONS:
Device: Oculus Quest — Virtual reality device to simulate specific exercises aimed at rehabilitating patients with musculoskeletal shoulder pathologies.
  Arms: Virtual reality-augmented shoulder rehabilitation

SUMMARY:
Malnutrition is a clinical syndrome defined by involuntary weight loss and/or a persistent imbalance between nutritional needs and intake, leading to functional decline. Its prevalence is particularly high among older adults-affecting about 17% of community-dwelling elders, 30% of those in rehabilitation settings, and between 20% and 60% of individuals in acute care environments. Malnutrition is therefore a common yet often underrecognized factor influencing health outcomes in geriatric populations.

Osteoarthritis (OA), a degenerative joint disease marked by the deterioration of articular cartilage, results in pain and reduced mobility. It affects approximately 9.6% of men and 18% of women over the age of 60. With global life expectancy rising and populations aging, OA is projected to become the fourth leading cause of disability by 2025. Joint replacement surgery provides significant relief for severe cases, and consequently, an increasing number of adults-averaging around 70 years of age-undergo elective joint replacement surgeries followed by rehabilitation for degenerative OA.

In this context, Virtual Reality (VR) technology is emerging as an innovative tool in rehabilitation. VR can create engaging, interactive environments that promote motor relearning by allowing clinicians to adjust practice intensity and provide real-time feedback. This adaptability enables personalized rehabilitation programs designed to enhance patient motivation and adherence. Preliminary studies have shown encouraging results, suggesting that VR-assisted therapy may improve motor recovery and functional outcomes, and its use in rehabilitation settings is rapidly expanding.

Previous research has identified a strong link between malnutrition and sarcopenia (loss of muscle mass) and reduced physical performance. However, findings remain inconsistent regarding how nutritional status influences functional recovery in elderly individuals undergoing rehabilitation. While some studies indicate a positive relationship between good nutrition and improved recovery, others suggest that nutritional status affects baseline functional capacity more than the rate or degree of functional improvement during rehabilitation.

It is also important to recognize that most available studies have focused on patients admitted for rehabilitation after hip fractures or stroke, conditions often associated with sudden functional decline. To date, only one known study has investigated elderly patients undergoing rehabilitation following hip or knee replacement surgery due to degenerative osteoarthritis. Interestingly, that study found a statistically significant positive association between nutritional status and functional recovery specifically in this subgroup-an association not observed among patients recovering from hip fractures or stroke.

Nonetheless, the study had limitations: nutritional status was measured using only the Mini Nutritional Assessment-Short Form (MNA-SF), and evaluation occurred post-surgery, without preoperative or long-term follow-up data. Moreover, there are no available data on rehabilitation outcomes for shoulder osteoarthritis, an increasingly common condition among older adults that significantly impacts autonomy in daily living.

Given these gaps, the current research aims to determine whether malnutrition modifies the effects of VR-enhanced shoulder rehabilitation after elective surgery on functional recovery-that is, the ability to perform activities of daily living (ADLs)-in frail elderly patients. The hypothesis is that poor nutritional status could reduce the benefits of intensive, technology-based rehabilitation, while adequate nutrition may enhance neuroplasticity, muscle strength, and overall recovery potential.

This investigation seeks to clarify three main aspects:

1. The prevalence and severity of malnutrition among elderly individuals undergoing elective surgery and subsequent VR-based rehabilitation.
2. The interaction between nutritional status and functional outcomes, examining whether malnutrition acts as an effect modifier or mediator in recovery trajectories.
3. The specific contribution of VR technology in improving rehabilitation adherence, motivation, and overall functional independence compared to conventional therapy.

By exploring the intersection between nutrition, aging, and digital rehabilitation, this research could help tailor multidisciplinary interventions that integrate nutritional management and advanced rehabilitation technologies. Such an approach may optimize recovery outcomes, reduce disability, and improve quality of life in frail older adults undergoing joint replacement or shoulder surgery due to osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 60 years old or older;
* Frailty defined according to the Clinical Frailty Scale (Cesari et al., 2018);
* Diagnosis of shoulder diseases with indication to elective surgery;

Exclusion Criteria:

* Diagnosis of rheumatic diseases;
* Shoulder fracture;
* Actual SARS-CoV-2 infection;
* Diagnosis of active cancer;
* Any contraindication to oral feeding;
* Malabsorptive diseases;
* Cognitive impairment (MMSE<18);
* Severe chronic diseases (heart failure NYHA III-IV, lung failure, renal failure);
* Any contraindication to rehabilitation;
* Rehabilitation duration ≤ 14 days;
* Inability to provide an informed consent;

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Malnutrition as effect modifier of the impact of shoulder rehabiliation | From enrollment to the end of rehabilitation treatment at 4 weeks
  "Absolute functional gain" (AFG), defined as the difference between the modified Barthel Index at the end of rehabilitation minus the modified Barthel Index before the rehabilitation (i.e. after surgery).

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Campus Bio-Medico, Rome, Rome, Italy